CLINICAL TRIAL: NCT07064122
Title: A Modular Phase I/II, Open-label, Multicentre Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of AZD2962, an IRAK4 Inhibitor, as Monotherapy and in Combination With Other Agents, in Participants With Haematologic Neoplasms
Brief Title: A Study of AZD2962, an IRAK4 Inhibitor (IRAK4 [a Body Protein] Blocker), in Participants With Haematologic Neoplasms (Blood Cancers)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7770C00001; 2025-520786-44 (Other: EU CT number); 172349 (Other: IND number)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Haematologic Neoplasms
Keywords: Interleukin-1 receptor associated kinase 4 (IRAK4) inhibitor; Modular study; Pharmacokinetics; Dose escalation
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Module 1- AZD2962 (Monotherapy) (Experimental): Participants with MDS and dysplastic CMML will receive AZD2962 as monotherapy in a dose escalation pattern.
  Interventions: Drug: AZD2962

INTERVENTIONS:
Drug: AZD2962 — AZD2962 will be administered orally once daily.

SUMMARY:
The purpose of the study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of AZD2962, an Interleukin-1 Receptor-Associated Kinase 4 (IRAK4) inhibitor, as monotherapy and in combination with other agents in participants with haematologic neoplasms.

DETAILED DESCRIPTION:
This is a modular study. In Module 1, the study will begin with a dose escalation of AZD2962 monotherapy in participants with myelodysplastic syndromes (MDS) and dysplastic chronic myelomonocytic leukemia (CMML).

Module 1 of the study will comprise of:

1. A Screening Period of maximum 21 days.
2. Treatment period with 28-day cycles where each patient will receive an oral dose of AZD2962 once daily, starting on Day 1, and will continue treatment until disease progression, unacceptable toxicity, or withdrawal.
3. Safety Follow-up period after 30 days after last dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with relapsed/refractory MDS or participants with relapsed/refractory dysplastic CMML, with peripheral blasts or bone marrow blasts < 20%, and who received one or more prior lines of therapy as per standard of care (or who exhausted locally available treatments including treatments for actionable mutations). Diagnosis must be histologically confirmed as per the WHO 2016 classification of myeloid neoplasms.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
3. Participants must have symptomatic disease that requires therapy and allows for objective efficacy assessments.
4. Willing to provide baseline bone marrow aspirate (or biopsy if dry-tap).
5. Contraceptive use by participants or participant partners should be consistent with local regulations and also comply with Clinical Study Protocol requirements.
6. All women of childbearing potential must have a negative serum pregnancy test result at Screening.

Key Exclusion Criteria:

1. Prior treatment with IRAK inhibitors or inhibitors of the inflammasome pathway.
2. Received any antineoplastic therapy (except hydroxyurea) within 15 days prior to first dose.
3. Received any strong or moderate Cytochrome P450 3A (CYP3A) inhibitors within 15 days prior to first dose.
4. Received major surgery within 28 days prior to first dose, or still recovering from surgery.
5. Received drugs that are known to prolong corrected QT interval (QTc) and with known risk of Torsades de Pointes, within 15 days prior to first dose.
6. Received immunosuppressive medications (including Graft-Versus-Host Disease prophylaxis) within 28 days prior to first dose, or within 15 days in the case of systemic steroids (doses exceeding 10 mg/day of prednisone or equivalent).
7. Received live attenuated vaccines within 28 days prior to first dose.
8. Active major bleeding event.
9. Any evidence of systemic disease, significant clinical disorder, or laboratory finding that make undesirable the participation in the study.

15. Mean resting corrected QT interval using Fridericia's formula (QTcF) > 450 ms obtained from triplicate Electrocardiograms (ECGs) and averaged, recorded within 5 minutes. In the presence of bundle branch block, QTcF > 470 ms is applicable.

16. History of intracranial bleeding within 6 months prior to first dose. 17. Active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism or excretion of oral therapy.

18. History of a prior non-haematologic neoplasm (with some exceptions). 19. Unresolved Grade > 2 toxicities from prior anticancer therapies (with some exceptions).

20. Concurrent enrolment in another clinical study (with some exceptions). 21. Known hypersensitivity to study intervention or its excipients.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) | From Cycle 1 Day 1 up to end of Cycle 1 (28 Days)
  A DLT is defined as an adverse event or abnormal laboratory value occurring during the DLT-evaluation period (first 28 days of treatment). This will be evaluated to assess the safety and tolerability and also to identify optimal biological dose (OBD) of AZD2962.
Number of participants with Adverse events (AEs) and serious AEs | Cycle 1 Day 1 up to safety follow-up (30 days after last dose) (Approximately 3 years)
  To assess the safety and tolerability of AZD2962 and also to identify OBD of AZD2962.
Duration of exposure | Cycle 1 Day 1 up to safety follow-up (30 days after last dose) (Approximately 3 years)
  To assess the safety and tolerability of AZD2962, and also to identify OBD of AZD2962.
Relative dose intensity | Cycle 1 Day 1 up to safety follow-up (30 days after last dose) (Approximately 3 years)
  To assess the safety and tolerability of AZD2962, and also to identify OBD of AZD2962.

SECONDARY OUTCOMES:
Percentage of participants with Objective response (OR) | First dose up to progression of disease (PD) or last evaluable assessment in the absence of progression, whichever comes first (Approximately 3 Years)
  For participants with MDS or CMML, OR is defined as the achievement of Best Overall Response (BOR) assessed by relevant criteria for the selected haematologic neoplasm. The OR will be assessed to estimate the efficacy of AZD2962.
Duration of response (DoR) | First documented response, up to the date of the first documented PD or study end, which ever comes first (Approximately 3 Years)
  The DoR is defined as the time from the date of first documented OR until date of first documented PD or death (by any cause in the absence of PD), regardless of discontinuation of study interventions or receiving another anticancer therapy. The DoR will be assessed to estimate the efficacy of AZD2962.
Time to Response (TTR) | First dose up to PD or last evaluable assessment, whichever comes first (Approximately 3 Years)
  The TTR is defined as the time between start of treatment and the date of documented confirmed objective response for the selected haematologic neoplasm. The TTR will be assessed to estimate the efficacy of AZD2962.
Overall Survival (OS) | First dose up to death due to any cause (Approximately 3 Years)
  The OS is defined as the time from the date of first dose until death due to any cause regardless of whether the participant withdraws from study therapy or receives another anti-cancer therapy. The OS will be assessed to estimate the efficacy of AZD2962.
Time to Progression to Acute myeloid leukaemia (AML) | First dose up to first diagnosis of AML (Approximately 3 Years)
  Time to progression to AML as per World Health Organization (WHO) 2016 is defined from the time of first dose until first diagnosis of AML, regardless of discontinuation of treatment or receiving another anti-cancer therapy. This will be assessed to estimate the efficacy of AZD2962.
Plasma concentration of AZD2962 | Cycle 1 Day 1 (each cycle is 28 days) up to end of the treatment (EoT) (Approximately 3 Years)
  To characterise the plasma concentration of AZD2962 as monotherapy.
Area under the concentration time curve (AUC). | Cycle 1 Day 1 (each cycle is 28 days) up to EoT (Approximately 3 Years)
  To characterise the pharmacokinetics (PK) AUC of AZD2962 as monotherapy.
Maximum plasma drug concentration (Cmax) | Cycle 1 Day 1 (each cycle is 28 days) up to EoT (Approximately 3 Years)
  To characterise the PK (Cmax) of AZD2962 as monotherapy.
Time to reach maximum concentration (tmax) | Cycle 1 Day 1 (each cycle is 28 days) up to EoT (Approximately 3 Years)
  To characterise the PK (tmax) of AZD2962 as monotherapy.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Heidelberg
  - Research Site, Melbourne
- Japan (2):
  - Research Site, Shinagawa-ku
  - Research Site, Yoshida-gun
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/